CLINICAL TRIAL: NCT06003452
Title: Retention Rate And Caries Prevention Of Giomer Based Sealant With And Without Pre-Treatment With Bioactive Glass Air Abrasion In Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, yomna sayed khallaf, lecturer at faculty of dentistry Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Fissure sealnt
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Dental Caries
Keywords: Fissure sealant; Bio-active glass; caries prevention
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Giomer Based Sealant Without Pre-Treatment With Bioactive Glass Air Abrasion (Active Comparator): giomer based fissure sealnt will be applied without surface treatment
  Interventions: Procedure: surface treatment with Bioactive Glass Air Abrasion
- Giomer Based Sealant With Pre-Treatment With Bioactive Glass Air Abrasion (Experimental): giomer based fissure sealnt will be applied after surface treatment With Bioactive Glass Air Abrasion
  Interventions: Procedure: surface treatment with Bioactive Glass Air Abrasion

INTERVENTIONS:
Procedure: surface treatment with Bioactive Glass Air Abrasion — giomer based fissure sealnt will be applied after surface treatment With Bioactive Glass Air Abrasion

SUMMARY:
Prevention of oral diseases is preferable to treatment and is the key method of achieving cost effectiveness for oral health improvement programs. Various preventive strategies for dental caries have been tried and are still being developed. The occlusal pits and fissures of posterior teeth are highly susceptible to caries because of the anatomy of pit and fissure surfaces, which favours stagnation of bacteria and substrates. Fissure sealing has been shown to be an evidence-based caries preventive method for protecting the occlusal surfaces against caries. Non- sealed teeth need to be restored approximately 50% more frequently compared to their sealed counterpart. Sealants are effective caries preventive agents as long as they remain bonded to teeth.

It has been proposed that sealants should be placed on both sound teeth and incipient non-cavitated carious lesions on permanent teeth of high caries risk patients in order to prevent the onset of caries and its progression. According to the American Dental Association Guidelines for the use of pit and fissure sealants, ICDAS II codes 0, 1 and 2 are recommended for sealant application.A variety of dental materials have been used as sealants using different application techniques. Their effectiveness depends on the formation of a complete seal and is increased by correct technique and moisture control, appropriate follow-up and resealing as necessary. Resin-based conventional sealants are preferred choice, however use of phosphoric acid demineralizes the enamel layer and have elongated treatment time and is more technique sensitive.

DETAILED DESCRIPTION:
It has been proposed that sealants should be placed on both sound teeth and incipient non-cavitated carious lesions on permanent teeth of high caries risk patients in order to prevent the onset of caries and its progression. According to the American Dental Association Guidelines for the use of pit and fissure sealants, ICDAS II codes 0, 1 and 2 are recommended for sealant application. A variety of dental materials have been used as sealants using different application techniques. Their effectiveness depends on the formation of a complete seal and is increased by correct technique and moisture control, appropriate follow-up and resealing as necessary. Resin-based conventional sealants are preferred choice, however use of phosphoric acid demineralizes the enamel layer and have elongated treatment time and is more technique sensitive3.

A new bioactive hybrid material (giomer) that combined the advantages of resin composites with glass ionomer cements has been introduced, it based on pre-reacted glass ionomer (PRG) filler technology in which fluoroaluminosilicate glass particles that have previously reacted with the polyacrylic acid were dispersed in resin. Giomer based pit and fissure sealant using self-etch primer eliminates phosphoric acid etch and rinse, thus conserving the enamel and reducing chair side time. However, retention of self-etch adhesive as compared to conventional sealants is questionable4.

A new method for sealant application using air- abrasive technology is less technique sensitive and allows for further cleaning of the grooves prior to sealant placement. The abrasive particles used in air abrasion effectively remove organic plug material from the grooves and allow for deeper penetration of the sealant material into the grooves5.

Aim of the study:

The aim of study is to evaluate retention rate and caries prevention of giomer based sealant with and without pre-treatment by bioactive glass air abrasion in young adults over one year

PICOTS:

(P) Patient/Population: Deep retentive fissures ( ICDAS 0,1,2) in second and third molars for 17-22 years old patients.

(I) Intervention: Giomer Based Sealant With Prior BioactiveGlass Air Abrasion. (C) Comparator: Giomer Based Sealant Without Prior Bioactive Glass Air Abrasion.

(O) Outcome:

Prioritization of Outcome

Outcome Method of Measurement (with reference)

Unit of Measurement

1. ry Outcome: Loss of retention Simonsen's criteria

   * Full retention (FR): The material was fully present on the occlusal surfaces
   * Partially lost (PL): The material was present, but as a result of either wear or loss of the material, part of a previously sealed pit or fissure, or both, was exposed
   * Totally lost (TL): No trace of the material was detected on the surface.
2. ry Outcomes Secondary Caries Modified USPHS criteria7 Alpha: Absence of the caries Charlie: Presence of the caries

(T) Time :- T0 :- Baseline T1:- 3 months Study Design: Two parallel arms randomized clinical trial. Study Framework: Superiority framework

Hypothesis:

The null hypothesis tested in this study is that there will be no difference either in the retention rate or caries prevention of giomer based sealant with and without treatment by bioactive glass air abrasion in young adults

Research question:

In deep retentive fissures, Will the use of bioactive glass air abrasion particles improve the retention rate and caries prevention of the giomer based sealant?

Methodology :

In Group 1: the self-etch primer (BeautiSealant Primer, Shofu, Japan) will be applied to the occlusal fissures with a fine micro brush. After waiting for 5 s, gently air blow for about 3 sec and then dry with stronger stream of air until a thin and uniform bonding layer is obtained. The giomer sealant. In Group 2: occlusal surface will be subjected to 5s of bioglass (AquaCare- Velopex International) , then sealant (BeautiSealant Paste, Shofu, Japan) will be applied as aforementioned steps and light-cured for 20 s. In both groups, the surfaces were checked with an explorer to ensure that no voids were present. The occlusion was checked and, if necessary, adjusted.

ELIGIBILITY:
Inclusion Criteria:

* Young adult Patients Aged 17-22.
* Good oral hygiene (plaque index score 0 or 1).
* Absence of abnormal occlusion habits (e.g. bruxism, nail biting, tooth clenching and mouth breathing).
* Patients approving to participate in the study.

Exclusion Criteria:

* Patients with known allergic or adverse reaction to the tested materials.
* Systematic disease that may affect participation.
* Xerostomic patients.

Ages: 17 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 96 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Loss of sealant's retention | 6 months
  Simonsen's criteria Full retention (FR) The material was fully present on the occlusal surfaces
  Partially lost (PL) The material was present, but as a result of either wear or loss of the material, part of a previously sealed pit or fissure, or both, was exposed
  - Totally lost (TL) No trace of the material was detected on the surface.

SECONDARY OUTCOMES:
Secondary Caries | 6 months
  Modified USPHS ( United States Public Health Service) criteria Alpha: Absence of the caries Charlie: Presence of the caries

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt